CLINICAL TRIAL: NCT03659994
Title: A Randomized, Double-blind, Clinical Trial to Compare the Effects of VitaBeard® on Facial Hair Growth in Healthy Adult Men
Brief Title: Effects of VitaBeard® on Facial Hair Growth in Healthy Adult Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Do Vitamins Inc. (Industry)
Collaborators: Nutrasource Pharmaceutical and Nutraceutical Services, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 1050-003-PRO-10072015
Record Dates: First submitted 2018-09-04; First posted 2018-09-06 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Healthy
Keywords: Facial Hair
MeSH Terms: interventions — Geritol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Vitabeard High Dose (Experimental): 3 capsules of multivitamin Vitabeard
  Interventions: Dietary Supplement: Multivitamin
- Vitabeard Mid-Dose (Experimental): 2 Capsules of multivitamin Vitabeard, 1 Capsule of Placebo
  Interventions: Dietary Supplement: Multivitamin
- Vitabeard Low-Dose (Experimental): 1 Capsule of multivitamin Vitabeard, 2 Capsules of Placebo
  Interventions: Dietary Supplement: Multivitamin
- Placebo (Placebo Comparator): 3 Capsules of Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Multivitamin — Vitabeard
  Arms: Vitabeard High Dose; Vitabeard Low-Dose; Vitabeard Mid-Dose
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine dose-dependent effects of Vitabeard on various parameters of facial hair growth.

DETAILED DESCRIPTION:
Primary and secondary assessments of efficacy will be made based on information obtained through hair measurements using Dermoscan and Trichoscan smart software. The device includes a camera handpiece with 5MP USB high resolution camera (Full HD) for standardized images and reproducible measurements. The Trichoscan smart software will be used for the measurement of hair parameters including hair count, hair density, hair width and hair length. Each subject will receive a permanent ink marking underneath the chin to standardize the location of assessments. Assessment periods over a 5 day period prior to baseline and a 5-day period at the end of the study. On the first day of each period, subjects will shave in the clinic and image is capture to demonstrate the clean shave of the area (Day 0), subjects do not shave for the following 5-days and images will be taken on Days 2 and 5 of each assessment period. Day 5 values will be used for comparing supplement effects (baseline to end of study, between groups). Day 2 will be used to calculate rate of growth during each assessment period, and will be used to compare supplement effects (baseline to end of study, between groups).

ELIGIBILITY:
Inclusion Criteria:

* Male aged 18 - 40 (inclusive)
* Healthy as determined from medical history
* Fitzpatrick skin type I-IV (See Appendix 1) with dark facial hair (brown or black)
* Non-smoker, or who quit smoking ≥6 months prior to visit 1
* Body mass index 18.0 - 29.9 kg/m2 (inclusive)
* Willing to avoid alcohol consumption 24 hours prior to the clinic visit and during the two 5-day assessment periods of facial hair growth
* Willing to maintain a stable body weight, activity level, sexual activity levels and dietary patterns, except for use of the study products, as directed
* Willing to maintain current outdoor activity amounts
* Willing to maintain current sexual activity level
* Willing to maintain current sleep habits
* Agrees to maintain current shaving habits during the study period with the exception of the assessment periods, during which participant agrees to avoid shaving
* Willing and able to provide consent for photographic release
* Willing and able to provide informed written consent

Exclusion Criteria:

* Individuals taking prescription or non-prescription health products that may affect the study endpoint in 6 months prior to visit 1 or during the study, such as hormone replacement therapy (testosterone, estrogen, progesterone, etc.), anabolic steroids, chemotherapy, intravenous or oral B vitamins, 5α-reductase inhibitors (e.g minoxidil, finasteride, etc.), medications with anti-androgenic properties (e.g. cyproterone, pironolacotne, ketoconazole, flutamide, bicalutamide), medications that can potentially cause hypertrichosis (e.g. ciclosporin, diazoxide, phenytoin, psoralens), oral glucocorticoids (inhaled glucocorticoids are permitted), lithium or phenothiazines, medications of known or suspected photoxocity (e.g., tetracyclines, thiazides, certain NSAIDs) and any other medications which, in the opinion of the investigator, may interfere with the performance of study assessments or place the subject at undue risk.
* Use of sulfonamides within 3 months prior to visit 1
* Unstable use (i.e. initiation or change in dose) medications for a thyroid condition within 3 months prior to visit 1
* Use of multivitamins within 2 weeks prior to visit 2a
* Use of Vitamin D containing supplements (≥500IU/day) within 4 weeks prior to visit 2a
* Use of Vitamin B7 (Biotin) containing supplements within 1 week prior to visit 2a
* Use of facial hair dyes (e.g. Just for Men®) in the previous 3 months and during the study
* Current use of depilatories, waxing, plucking or bleaching or current or prior use at any time of laser hair removal on the target test or surrounding area to an extent which, in the opinion of the investigator, may interfere with the performance of the study assessments
* Very little contrast between hair color and scalp (e.g., fair-haired with an extremely pale skin color)
* Use of any weight-loss programs or weight-loss medications (prescription or over-the counter) including, but not limited to, lipase inhibitors, within 6 months prior to visit 1 and throughout the study
* Individuals with an outdoor occupation (e.g. landscaper, surveyor, outdoor construction, etc.)
* Active skin diseases (e.g. eczema, atopic dermatitis, psoriasis, skin cancer, sun damaged skin with actinic keratosis, on facial/chin area)
* Damaged skin in or around test site including sunburn, uneven skin tones, tattoos, scars or other disfiguration of the test site
* Routine high dosage use of anti-inflammatory medications (such as aspirin, ibuprofen, corticosteroids, etc), immunosuppressive drugs or antihistamine medications. Steroid nose drops and/or eye drops are permitted. Two 81mg or one 325mg aspirin per day is also permitted.
* Use of topical drugs on the face or underneath chin area
* History of disorders affecting biotin metabolism (e.g. holocarboxylase synthetase (HCS) deficiency, biotinidase deficiency, biotin-responsive basal ganglia disease, multiple carboxylase deficiency)
* Presence of major diseases such as diabetes, gastrointestinal, endocrine, cardiovascular, renal, or liver disease
* History of neurological disease (e.g. Parkinson's disease, stroke, traumatic brain injury, etc.)
* History of cancer in the past 5 years
* Uncontrolled hypertension defined as a seated resting systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg
* Abnormal laboratory test results of clinical significance, including, but not limited to ALT or AST ≥1.5X the upper limit of normal at screening (Visit 1)
* Presence or history (past 6 months) of alcohol or drug abuse; alcohol use of >2 standard alcoholic drinks per day
* Participant has a known allergy or intolerance to any of the ingredients in the test product or placebo
* Participant is unwilling or unable to abide by the requirements of the protocol
* Any condition that would interfere with the participant's ability to comply with study instructions, might confound the interpretation of the study, or put the participant at risk
* Participant has taken an investigational medicine or has participated in a research study within 30 days prior to first study visit

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Rate of Facial Hair Growth | 33 Days
  Rate of hair growth will be determined as the change in length of hair from day 2 to day 5 of each assessment period (beginning of study and end of study) divided by the number of days. Hair length was obtained using Trichoscan software and images captured with Dermoscan

SECONDARY OUTCOMES:
Facial hair density | 33 days
  Determined as the number of hairs in a standardized area calculated automatically by Trichoscan software and images captured with Dermoscan
Facial hair strand thickness | 33 days
  Hair width determined automatically using Trichoscan software and images captured with Dermoscan

CONTACTS AND LOCATIONS:
Locations (1):
- Nutrasource, Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No